CLINICAL TRIAL: NCT04945915
Title: Prediction of Postoperative Pulmonary Complications Using Damage-associated Molecular Patterns in Adult Cardiac Surgery
Brief Title: Prediction of PPC Using DAMPs in Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2018-139
Record Dates: First submitted 2021-06-16; First posted 2021-06-30 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery; Damage-associated Molecular Patterns
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected four times in total, and 7 ml of blood was collected after induction of anesthesia (T1), 90 minutes after CPB (T2), immediately after weaning from CPB (T3), and on the first day after surgery (T4). It was placed in a serum-separating tube and then centrifuged. Enzyme-linked immune sorbent assay is performed to measure the concentration of heparan sulfate (HS) and high mobility group box 1 (HMGB1) using HS ELISA kit (Finetest, EH4010) and HMGB1 ELISA kit (Solarbio, SEKH-0409), respectively. use.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — There was no intervention because this reasearch is observational study.

SUMMARY:
DAMPs (damage associated molecular patterns) are endogenous molecules that are expressed by cell stress or cell damage and play an important role in tissue (or host) defense and repair by activating the innate immune system. This is not the case with infections or injuries. Briefly, it starts when the immune system is activated by a receptor that recognizes a damage pattern, and it is a generic term for continuous responses by endogenous molecules expressed in this process. Recently, immuno-cancer drugs for cancer treatment by applying this immune response are also emerging. In cardiac surgery using cardiopulmonary bypass (CPB), there are more deleterious effects and adverse effects caused by using CPB than the surgery itself. There are several studies that have revealed the association between DAMPs and the degree of complications by approaching them from the point of view of tissue damage caused by the use of CPB. Therefore, we intend to investigate the changes in DMAPs over time during, and after cardiac surgery and the differences in DAMPs according to the presence or absence of postoperative pulmonary complications.

DETAILED DESCRIPTION:
DAMPs (damage-associated molecular patterns) are endogenous molecules expressed as a result of cell stress or damage. They play a crucial role in tissue or host defense and repair by activating the innate immune system. This differs from cases of infections or injuries. In a nutshell, the process begins when the immune system is triggered by a receptor that recognizes a damage pattern. DAMPs is a broad term encompassing continuous responses by endogenous molecules expressed during this process. More recently, there has been a growing focus on using this immune response for cancer treatment through immuno-cancer drugs. In cardiac surgery using cardiopulmonary bypass (CPB), various types of damage occur, including intravascular cannulation, exposure to the surface of the bypass circuit, ischemia-reperfusion injury, and surgical injury (operative trauma). During this process, the expression of pro-inflammatory cytokines and DAMPs (damage-associated molecular patterns) takes place. This leads to a response similar to sterile systemic inflammatory response syndrome (SIRS). As a result of this process, patients become more vulnerable to post-surgery infections or remote organ failure due to immune suppression.

Several studies have explored the link between DAMPs and the extent of complications by assessing tissue damage resulting from CPB usage. However, there is no study on the relationship between the occurrence of pulmonary complications and DAMPs in cardiac surgery, and therefore the authors aimed to determine changes in DMAPs over time during, and after cardiac surgery and the differences in DAMPs according to the presence or absence of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 20 years of age
* Patients undergoing cardiac surgery using cardiopulmonary bypass (CPB)

Exclusion Criteria:

* pregnant women and minors
* the patients who required mechanical life support as follows due to unstable vital signs after CPB weaning, ECMO (extracorporeal membrane oxygenation) IABP (intra-aortic balloon pump)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery using cardiopulmonary bypass (CPB)
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Concentration of heparan sulfate (HS) | the day after surgery, up to 48hours
  blood sampling before CPB application, 90 minutes after CPB application, after CPB weaning, the day after surgery
Concentration of high mobility group box 1 (HMGB1) | the day after surgery, up to 48hours
  blood sampling before CPB application, 90 minutes after CPB application, after CPB weaning, the day after surgery

SECONDARY OUTCOMES:
Postoperative complication | during admission, up to 22 days
  By evaluating clinical recovery through the presence or absence of postoperative complications, the relationship between the concentration of DAMPs and the patient's clinical prognosis is investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea